CLINICAL TRIAL: NCT06439576
Title: China Faricimab Real World Evidence: Evaluation of Faricimab Effectiveness, Safety and Treatment Pattern, in Diabetic Macular Edema, Retinal Vein Occlusion and Neovascular Age-Related Macular Degeneration: The Farseeing Study
Brief Title: Real World Evidence in China: Faricimab Use in Diabetic Macular Edema, Retinal Vein Occlusion, and Neovascular Age-Related Macular Degeneration (The Farseeing Study)
Status: Recruiting | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Shanghai Roche Pharmaceutical Co., Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: ML45401
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Diabetic Macular Edema; Neovascular Age-related Macular Degeneration; Retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — faricimab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1: Patients with nAMD
  Interventions: Drug: Faricimab
- Cohort 2: Patients with DME
  Interventions: Drug: Faricimab
- Cohort 3: Patients with RVO
  Interventions: Drug: Faricimab

INTERVENTIONS:
Drug: Faricimab — The dosing and treatment duration of the studied medicinal product is at the discretion of the physician in accordance with clinical practice and labeling in China.
  Other Names: VABYSMO®

SUMMARY:
The Farseeing Study will explore long-term effectiveness, safety, and treatment patterns among patients being treated with faricimab in real-world, routine clinical practice in China. It is a primary data collection, non-interventional, prospective and retrospective, multi-center study designed to collect real-world, long-term data to gain clinical evidence on faricimab, by observing cohorts of patients with neovascular age-related macular degeneration (nAMD), diabetic macular edema (DME), and retinal vein occlusion (RVO) who are receiving treatment with faricimab.

ELIGIBILITY:
Inclusion Criteria:

1. Have signed the informed consent
2. Female and male Chinese patients, who had been diagnosed with nAMD, DME, or RVO by CFP, OCT, FFA, ICGA, or OCTA
3. ≥50 years old for patients with nAMD, ≥18 years old both for patients with DME and RVO, at the time of signing informed consent (or the first administration of faricimab, whichever occurs first)
4. Patients for whom the decision to receive treatment with faricimab is made prior to and independent from study participation
5. Patients have received at least one faricimab treatment (the first dose) in the study eye

Exclusion Criteria:

1. Patients not receiving treatment for nAMD/DME/RVO with faricimab according to the standard of care and in line with the current summary of product characteristics (SPC) / labeling in China
2. Active ocular inflammation or suspected / active ocular infection in either eye
3. Received any other anti-VEGF treatment after faricimab
4. Received any steroid treatment within 6 months (180 days) before the first faricimab treatment in the study eye
5. Any participation in any other clinical trials currently
6. Patients could not provide the clinical data (visual acuity and OCT images) within 2 weeks (14 days) before receiving the initial faricimab injection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will recruit patients who are naïve to anti-VEGF therapy in the study eye and those who have previously been treated with anti-VEGF therapy in the study eye. Study participation of patients previously treated with other anti-VEGF agents will be capped at a maximum of 40% of each indication enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2027-11-15 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Acuity from Baseline at Month 12 | Baseline and Month 12
  Visual acuity will be collected as measured per local practice and then will be converted to the approximate ETDRS letter score.

SECONDARY OUTCOMES:
Visual Acuity Over Time | Baseline, Months 3, 6, 9, 12, 18, and 24
Change in Visual Acuity from Baseline Over Time | Baseline, Months 3, 6, 9, 18, and 24
Central Subfield Thickness Over Time | Baseline, Months 3, 6, 9, 12, 18, and 24
Change in Central Subfield Thickness from Baseline Over Time | Baseline, Months 3, 6, 9, 12, 18, and 24
Percentage of Eyes on Each Treatment Regimen (Fixed, Treat-and-Extend, As Needed, or Other) | From Baseline to Month 24
Number of Treatments per Year | Months 12 and 24
Percentage of Eyes with Treatment Switch by Reason for Switch Over Time | Months 3, 6, 9, 12, 18, and 24
Percentage of Eyes with Treatment Regimen Switch (Fixed, Treat-and-Extend, As Needed, or Other) by Reason for Switch Over Time | Months 3, 6, 9, 12, 18, and 24
Total Number of Visits per Year | Months 12 and 24
Number of Visits With or Without Treatment per Year | Months 12 and 24
Time Interval Between Treatments per Year | Months 12 and 24
Percentage of Eyes Treated with Ocular Concomitant Medications or Therapy by Type and Frequency During the Study | From Baseline until end of study (up to 3.5 years)
Number of Participants Lost to Follow-Up More Than 6 Months at Months 12, 18, and 24 | Months 12, 18, and 24
Percentage of Eyes According to the Last Treatment Interval at Months 3, 6, 12, 18, and 24 | Months 3, 6, 12, 18, and 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (41):
- China (41):
  - Joint Shantou International Eye Center, Shantou, Guangdong
  - The First Affiliated Hospital of Henan UN of Science and Technology, Luoyang, Henan
  - Taihe Hospital of Shiyan, Shiyan, Hubei
  - Xuzhou No.1 Peoples Hospital, Xuzhou, Jiangsu
  - Fushun Eye Hospital, Fushun, Liaoning
  - Panjin Central Hospital, Panjin, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Affiliated Hospital of Shandong Second Medical University, Weifang, Shandong
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - The First People's Hospital of Chengdu, Chengdu, Sichuan
  - The First People's Hospital of Kashgar, Kashgar, Xinjiang Uygur
  - The First People's Hospital of Yunnan Province, Kunming, Yun'nan
  - Jinhua municipal central hospital, Jinhua, Zhejiang
  - Peking University People's Hospital, Beijing
  - Sichuan Provincial People's Hospital, Chengdu
  - People's Hospital of Dingzhou, Dingzhou
  - Dongyang People's Hospital, Dongyang
  - Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou
  - Guizhou Provincial People's Hospital, Guiyang
  - Eye Hospital of Shandong First Medical University, Jinan
  - The First Affiliated Hospital of Lanzhou University, Lanzhou
  - The Affiliated Hospital of Southwest Medical University, Zhongshan Campus, Luzhou
  - Jiangsu Province Hospital (the First Affiliated Hospital With Nanjing Medical University), Nanjing
  - The People?s Hospital of Guangxi Zhuang Autonomous Region, Nanning
  - Qingdao Eye Hospital of Shandong First Medical University, Qingdao
  - Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai Tenth People's Hospital, Shanghai
  - Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - Shanghai Zhoupu Hospital, Shanghai
  - Shenyang Fourth People's Hospital, Shenyang
  - Shenzhen Eye Hospital, Shenzhen
  - Hebei People's Hospital, Shijiazhuang
  - Shanxi Bethune Hospital, Taiyuan
  - Tianjin Eye Hospital, Tianjin
  - Eye Hospital, Wenzhou Medical University, Wenzhou
  - Xiehe Hospital, Tongji Medical College Huazhong University of Science & Technology, Wuhan
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Xiamen Eye Center Of Xiamen University, Xiamen
  - Hebei Eye Hospital, Xingtai
  - Henan Provincial Eye Hosptial, Zhengzhou
  - Affiliated Hospital of Zunyi Medical University, Zunyi

IPD SHARING:
Plan to Share IPD: No